CLINICAL TRIAL: NCT03128268
Title: THE EFFECTIVENESS OF 4D IMAGE ACQUISITION AND POST-PROCESSING WITH VIOS WORKS: A Phase Design Prospective Clinical Trial to Assess 4D Software Produced by GE and Arterys for Evaluating Cardiac Disease.
Brief Title: The Effectiveness of 4D Image Acquisition and Post-processing With Vios Works
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: GE Healthcare (Industry); Arterys, Inc. (Unknown)
Responsible Party: Principal Investigator, Michael Poon, Chief, Non-invasive Cardiac Imaging, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-845-LHH
Record Dates: First submitted 2017-04-03; First posted 2017-04-25 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: Each participant will receive tradition 2D Cardiac imaging as ordered per standard of care. Then, the participant will receive a 4D image, requiring 6 to 10 additional minutes in the MRI scanner. The 2D and 4D images will be interpreted by readers blinded to the results of the alternate modality. Inter- and intra-reader reliability will be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- All Enrollees (Experimental): Intervention: Diagnostic test
  All enrollees will receive a 4D MRI as a research intervention using imaging software for 4 dimensional images for Cardiac MRI
  Interventions: Device: Imaging software for 4 dimensional images for Cardiac MRI

INTERVENTIONS:
Device: Imaging software for 4 dimensional images for Cardiac MRI — All enrollees will receive Cardiac MRI scans using Imaging software for 4 dimensional images for Cardiac MRI

SUMMARY:
This study aims to evaluate the effectiveness of 4D image acquisition and post-processing with Vios Works for the evaluation of 3D images acquired on GE Magnetic Resonance Imaging scanners. Specifically, the investigators propose to evaluate the following:

1. Image acquisition time using traditional 2D and new 4D processing techniques;
2. Image quality for 2D and 4D processing techniques subjectively
3. Post-processing time for the two techniques.
4. Correlation of overall Left ventricular and right ventricular volumes and functions and aortic and pulmonic flow studies using the two techniques.
5. The study will monitor any changes in patient diagnoses or treatment resulting from any differences in interpretations between the two processes.

DETAILED DESCRIPTION:
Traditional scanning and post-processing of 2D Cardiac Magnetic Resonance images (CMRI) is highly technical and time consuming, with many exams requiring one to two hours to complete. In addition, performance of 2D scans often requires expert technologists working closely with the clinician imaging expert. These factors limit the general clinical utility of current generation cardiac MRI.

In order to address these factors, many researchers began to explore the use of 4D image acquisition and post processing to shorten exam time. These researchers have documented success at these efforts but, to the best of the current investigators' knowledge, such advanced imaging acquisition and post-processing systems are not readily commercially available in the US.

Recently GE teamed with Vios-Works for MRI to provide a cloud-based visualization platform for 4D MRI that provides quantitative and structured reporting in the post processing environment that makes use of advance MR imaging acquisition techniques. The images can be accessed by the interpreter and reviewed and manipulated in order to assess cardiac function and flow retrospectively, which, prior to this innovation, only has been available for computed tomography (CT) generated images.

This investigative team hypothesizes that the use of 4D imaging will result in reduced time for acquisition (approximately 6 minutes as opposed to 1 hour), and improvement of diagnostic capability.

Images will be acquired using the current standard 2D acquisition protocol for routine clinical cardiac MRI. A repeat acquisition will be completed using the new protocol for 4D imaging acquisition. This will require that patient exams be extended in length by six minutes for those enrolled in the study. The investigators will evaluate the image quality of the two techniques and grade them according to a scale of 1 to 3 with 1 being excellent cardiac borders easily identified; 2 - acceptable: cardiac borders acceptably identified; and 3, non-diagnostic. The investigators will specifically focus on the evaluation of cardiac function of both right and left ventricular function as well as flow analysis of both the aortic and pulmonic valves.

For each method, technician time and MD time will be collected. The exam will go through post processing for standard 2D, following by the new 4D post processing technique. Time for post processing will be collected. All subjects who agree will receive both a 2D and a 4D MRI. The investigators will evaluate inter and intra reader reliability by having all readers read the first 15 exams, and then read them a second time after two weeks in a different order Readers showing variation in performance will be retrained on interpretation of 4D MRI before reading scans for the study.

Once readers have been trained, the study will require that all 2D and 4D exams be read by two readers. The exams will be assigned randomly to readers using the Biostatistician Office random assignment services.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* with a valid prescription for Cardiac MRI for the following: Congenital heart disease/Shunts, Valvular heart disease, Pulmonary Hypertension, Aortic Disease, Hypertrophic Cardiomyopathy (HCM)
* receiving Standard of Care services at the MRI Center
* consent to participate in the 4D trial

Exclusion Criteria:

Patients with any of the following will be excluded:

* Pacemaker or ICD implanted
* ICDs implanted
* Temporary Pacemakers (e.g. transvenous temporary wires)
* Leads that are abandoned (capped or retained leads not attached to device)
* Non-transvenous leads (e.g. epicardial leads)
* Leads that have no fixation (e.g. floating leads)
* A lead that is known to be fractured
* Any other metallic objects that, in the opinion of the safety officer would compromise patient safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
2D imaging findings and medical diagnoses resulting from images. | Investigators are expected to interpret the 2D images in one sitting requiring 15 minutes to three hours, depending on exam complexity. The investigator will complete the scan review within 1 day to 1 month of the exam date.
  Investigators will count the number of study outcomes documented that are related to patient treatment.
4D imaging findings and medical diagnoses resulting from images. | Investigators are expected to interpret the 4D images in one sitting requiring 15 minutes to three hours, depending on exam complexity. The investigator will complete the scan review within 1 day to 1 month of the exam date.
  Investigators will count the number of study outcomes documented that are related to patient treatment.

SECONDARY OUTCOMES:
2D Time to scan acquisition | The 2D scan time will be from the time the 2D patient scan starts to the time the 2D patient scan ends. These will be measured on the patient's scheduled scan date.
  Investigators will document time to acquire 2D image.
Time to 2D scan interpretation | The time required for the reader to interpret scan for 2D and to document results. Within one month of scan completion. Reader is expected to interpret each scan in 1 to 3 hours.
  Time to interpret 2-D scan interpretation will be from the time the reader starts reading the 2D scan until the time the reader finishes reading the 2D scan.
Intra-reader reliability | The reader will record all findings from each scan immediately upon completion of scan interpretation. Findings should be recorded within a month of the exam.
  Each reader will read each scan assigned on two different dates. The reader will be blind to identity of scan. The two readings will be compared for consistency.
Image quality | The reader will record an image score for each exam during interpretation of the scan. The reader will record an image score within one month of scan completion date.
  Overall measure of all scan image quality based on standard quality assessment protocol definitions.
2D patient recommended treatments | The reader will recommend follow-up patient care for each patient based upon completion of the exam interpretation. The reader will record all recommendations within one month of the exam.
  The reader will document recommendations for patient treatment based on 2D imaging results
90 day follow up | The interviewer will contact patients with a target date of 90 to 120 days after the exam to obtain the followup information via telephone.
  Describe patient follow-up. The interviewer will record the patient follow up by interviewing the patient within 90 to 120 days of the scan and asking what follow up was taken; and by medical record review. Follow up will be recorded and will be compared to recommended follow up.
4D Time to scan acquisition | The 4D scan time will be from the time the 4D patient scan starts to the time the 4D patient scan ends. These will be measured on the patients scheduled scan date.
  Investigators will document time to acquire 4D image
Time to 4D scan interpretation | The time required for the reader to interpret scan for 4D and to document results. Within one month of scan completion. Reader is expected to interpret each scan in 1 to 3 hours.
  Time to interpret 4D scan interpretation will be from the time the reader starts reading the 4D scan until the time the reader finishes reading the 4D scan.
Inter-reader reliability | The reader will record all findings from each scan immediately upon completion of scan interpretation. Findings should be recorded within a month of the exam.
  Two readers will read each scan. The readers will be blind to identity of scan. the reader will not know the results reported by the second reader. The two readings will be compared for consistency.
4D patient recommended treatments | The reader will recommend follow-up patient care for each patient based upon completion of the exam interpretation. The reader will record all recommendations within one month of the exam.
  The reader will document recommendations for patient treatment based on 4D imaging results

CONTACTS AND LOCATIONS:
Overall Officials: Michael Poon, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health Imaging at Greenwich Village: a Division of Lenox Hill Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Okada RD, Lim YL, Rothendler J, Boucher CA, Block PC, Pohost GM. Split dose thallium-201 dipyridamole imaging: a new technique for obtaining thallium images before and immediately after an intervention. J Am Coll Cardiol. 1983 May;1(5):1302-10. doi: 10.1016/s0735-1097(83)80144-2. No abstract available. PMID 6833669
- [Background] Vasanawala SS, Hanneman K, Alley MT, Hsiao A. Congenital heart disease assessment with 4D flow MRI. J Magn Reson Imaging. 2015 Oct;42(4):870-86. doi: 10.1002/jmri.24856. Epub 2015 Feb 24. PMID 25708923
- [Background] Hsiao A, Alley MT, Massaband P, Herfkens RJ, Chan FP, Vasanawala SS. Improved cardiovascular flow quantification with time-resolved volumetric phase-contrast MRI. Pediatr Radiol. 2011 Jun;41(6):711-20. doi: 10.1007/s00247-010-1932-z. Epub 2011 Jan 11. PMID 21221566
- [Background] Hsiao A, Lustig M, Alley MT, Murphy M, Chan FP, Herfkens RJ, Vasanawala SS. Rapid pediatric cardiac assessment of flow and ventricular volume with compressed sensing parallel imaging volumetric cine phase-contrast MRI. AJR Am J Roentgenol. 2012 Mar;198(3):W250-9. doi: 10.2214/AJR.11.6969. PMID 22358022
- [Background] Hsiao A, Lustig M, Alley MT, Murphy MJ, Vasanawala SS. Evaluation of valvular insufficiency and shunts with parallel-imaging compressed-sensing 4D phase-contrast MR imaging with stereoscopic 3D velocity-fusion volume-rendered visualization. Radiology. 2012 Oct;265(1):87-95. doi: 10.1148/radiol.12120055. Epub 2012 Aug 24. PMID 22923717
- [Background] Uretsky S, Gillam L, Lang R, Chaudhry FA, Argulian E, Supariwala A, Gurram S, Jain K, Subero M, Jang JJ, Cohen R, Wolff SD. Discordance between echocardiography and MRI in the assessment of mitral regurgitation severity: a prospective multicenter trial. J Am Coll Cardiol. 2015 Mar 24;65(11):1078-88. doi: 10.1016/j.jacc.2014.12.047. PMID 25790878
- [Background] Dyverfeldt P, Bissell M, Barker AJ, Bolger AF, Carlhall CJ, Ebbers T, Francios CJ, Frydrychowicz A, Geiger J, Giese D, Hope MD, Kilner PJ, Kozerke S, Myerson S, Neubauer S, Wieben O, Markl M. 4D flow cardiovascular magnetic resonance consensus statement. J Cardiovasc Magn Reson. 2015 Aug 10;17(1):72. doi: 10.1186/s12968-015-0174-5. PMID 26257141